CLINICAL TRIAL: NCT04517747
Title: A Pilot Study of Ramucirumab Beyond Progression Plus TAS-102 in Patients With Advanced or Metastatic Adenocarcinoma of the Stomach or the Gastroesophageal Junction, After Treatment Failure on a Ramucirumab Based Therapy
Brief Title: Ramucirumab Plus TAS-102 in Patients With Advanced or Metastatic Gastric Adenocarcinoma or the Gastroesophageal Junction
Acronym: RE-ExPEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RE-ExPEL
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Gastric Adenocarcinoma; Metastatic Adenocarcinoma of the Gastroesophageal Junction
MeSH Terms: interventions — Ramucirumab; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ramucirumab plus TAS-102 (Experimental): Ramucirumab 8 mg/kg i.v. on day 1 and day 15 of a 28-day cycle and TAS-102 35 mg/m2/dose p.o. twice daily on days 1 to 5 and days 8 to 12 of a 28-day cycle Each cycle will be repeated after 28 days (from day 1) for a maximum of 4 cycles.
  Interventions: Drug: Ramucirumab; Drug: TAS 102

INTERVENTIONS:
Drug: Ramucirumab — chemotherapy i.v.
  Other Names: Cyramza
Drug: TAS 102 — p.o. twice daily
  Other Names: Lonsurf

SUMMARY:
The objective of this study is to determine whether a combination of ramucirumab, beyond progression after a SOC 2nd line ramucirumab based pre-treatment (Ram beyond progression) in patients with locally advanced or metastatic adenocarcinoma, plus TAS-102 shows good tolerability without safety issues regarding the serious adverse event rate of any cause, and whether the combination shows positive signals regarding efficacy in the secondary endpoints (e.g. prolongation of progression-free survival of TAS-102 plus ramucirumab compared with TAS-102 monotherapy - historical data according to TAGS trial).

DETAILED DESCRIPTION:
This is an interventional, prospective, non-randomized, open-label, multicenter single-arm pilot study of ramucirumab plus TAS-102 in patients with advanced or metastatic adenocarcinoma of the stomach or the gastroesophageal junction, after treatment failure on a ramucirumab based therapy.

A total number of 20 patients will be enrolled. Potential study participants will be assessed for eligibility during one or several screening visits. The patient has to provide a signed informed consent form prior to any study-specific screening evaluations. Once the patient provides a signed informed consent form and eligibility is confirmed (all inclusion/exclusion criteria have been verified), the patient can be enrolled.

All screening procedures must be completed during the 14-day screening period. All patients must have had disease status confirmed as per CT or MRI scan of the tumor(s) within ≤ 4 weeks prior to the first dose. Other screening assessments include blood sampling, performance status (ECOG) and ECG according to clinical routine. Study treatment will be continued until progression or intolerable toxicity, but for a maximum of 4 months. Further treatment after progression will be at the investigator's discretion.

Tumor assessment will be performed according to clinical routine at screening and every 8 weeks (±7 days) during the treatment phase of the study and every 12 weeks (±14 days) during follow-up.

The expected duration of the active study phase (FPI - LPO) is 18 months. The active phase per individual patient is approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Men or women* ≥ 18 years of age. Patients of reproductive age must be prepared to use a suitable contraceptive method during the study and up to 6 months after the end of treatment. A suitable method of contraception is defined as surgical sterilization (e.g. bilateral fallopian tube ligation, vasectomy), hormonal contraception (implantable, patch, oral), and double barrier methods (each two-fold combination of intrauterine pessary, condom for men, or women with spermicidal gel, diaphragm, contraceptive sponge, cervical cap). Women of child-bearing potential must have a negative pregnancy test within the last 7 days prior to the start of study therapy.

   *There is no data that indicates a specific gender distribution. Therefore, patients are included regardless of their gender.
3. Histologically proven adenocarcinoma of the stomach, including adenocarcinoma of the gastroesophageal junction (note: previous histological assessment during disease history of patient sufficient, current biopsy during screening for this trial is not mandatory)
4. Documented, objective, radiological or clinical progression of the disease during or within 4-6 weeks after the last dose of a ramucirumab based second-line therapy (ramucirumab monotherapy or a combination of ramucirumab + paclitaxel, respectively ramucirumab + FOLFIRI).
5. Measurable or non-measurable but evaluable disease.
6. ECOG Performance status 0-2.
7. Life expectancy > 8 weeks.
8. Appropriate haematological, hepatic and renal function:

   1. Absolute number of neutrophils (ANC) ≥ 1.5 x 10^9/L
   2. Platelets ≥ 100 x 10^9/L
   3. Hemoglobin ≥ 9 g/dL (5.58 mmol/L)
   4. Total bilirubin ≤ 1.5 times the upper limit of normal (UNL)
   5. AST (SGOT) and ALT (SGPT) ≤ 2.5 x UNL without existing liver metastases, or ≤ 5 x UNL in the presence of liver metastases; AP ≤ 5 x UNL
9. Serum creatinine ≤ 1.5 x UNL or creatinine clearance (measured by 24h urine) ≥ 40 mL / min (i.e. if the serum creatinine level is > 1.5 x UNL, then a 24h urine test must be performed to check the creatinine clearance to be determined). Protein level in urine ≤ 1+ by dipstick analysis or routine urine measurement (if the dipstick analysis or the routine test ≥ 2+, a subsequent 24h urine protein measurement must show a value of < 1000mg of protein within 24h of participation to ensure the study.
10. Adequate coagulability, as determined by the International Normalized Ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT) ≤ 5 seconds above the UNL (unless anti-coagulation therapy has been given). Patients receiving warfarin / phenoprocoumon must be switched to low molecular weight heparin and must have a stable coagulation profile before starting study-specific therapy.
11. Subject is willing and able to comply with the protocol (including contraceptive measures) for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Presence of tumors other than adenocarcinomas (e.g., leiomyosarcoma, lymphoma) or a secondary tumor other than squamous or basal cell carcinomas of the skin or in situ carcinomas of the cervix which have been effectively treated. The sponsor decides to include patients who have received curative treatment and have been disease-free for at least 5 years.
2. Squamous cell carcinoma of the stomach or gastroesophageal junction.
3. Simultaneous, ongoing, systemic immunotherapy, chemotherapy, or hormone therapy not described in the study protocol.
4. Simultaneous treatment with a different anti-cancer therapy other than that provided for in the study (excluding palliative radiotherapy for symptom control).
5. The patient is receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted
6. The patient has undergone major surgery within the last 28 days prior to the start of study-specific therapy or has undergone minor surgery within the last 7 days prior to the start of study therapy. The patient had subcutaneous venous access within the last 7 days prior to the start of the study-specific therapy. The patient plans to undergo major surgery while participating in the clinical trial.
7. Gastrointestinal bleeding grade 3-4 within the last 3 months prior to enrollment in the study.
8. History of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other clinically important thromboembolic event during the last 3 months prior to the start of study-specific therapy (thrombosis caused by venous ports, catheters, or superficial venous thrombosis are not considered "clinically meaningful").
9. Stage B cirrhosis according to Child-Pugh criteria (or worse) or cirrhosis (of any grade) with a history of hepatic encephalopathy or clinically significant ascites resulting from cirrhosis. Clinically significant ascites is defined as ascites resulting from cirrhosis requiring diuretics or paracentesis.
10. Known brain or leptomeningeal metastases.
11. Known allergic / hypersensitive reactions to at least one of the treatment components.
12. Other serious illnesses or medical ailments within the last 12 months prior to the start of the study.
13. Any arterial thromboembolic event which includes, but is not limited to, the following: myocardial infarction, transient ischemic attack, cerebrovascular insult, unstable angina within the last 6 months prior to the initiation of study therapy.
14. Uncontrolled or under-adjusted hypertension (> 160 mmHg systolic or > 100 mmHg diastolic hypertension for more than 4 weeks) despite standard medical treatment.
15. Presence of an active, uncontrollable infection.
16. Chronic inflammatory bowel disease.
17. Active disseminated intravascular coagulation.
18. Any other serious concomitant or medical condition that, in the opinion of the investigator, presents a high risk of complications to the patient or reduces the likelihood of clinical effect.
19. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
20. History of gastrointestinal perforation / fistula (within the last 6 months prior to the start of study-specific therapy) or presence of risk factors favoring perforation.
21. Serious or non-healing wounds, ulcers, or broken bones within the last 28 days prior to the start of study-specific therapy.
22. The patient is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Tolerability and toxicity: rate of serious adverse events (SAEs) of any cause | Frist Treatment until 30 days after end of treatment, up to 5 months
  The primary endpoint of the study is tolerability and toxicity, defined by the rate of serious adverse events (SAEs) of any cause according to CTCAE v5.0

SECONDARY OUTCOMES:
Rate of treatment-related AEs and SAE | Frist Treatment until 30 days after end of treatment, up to 5 months
  Rate of treatment-related AEs and SAEs according to CTCAE v5.0
Adverse events for neutropenia | Frist Treatment until 30 days after end of treatment, up to 5 months
  Rate of grade 3 or worse adverse events for neutropenia
Adverse events for anemia | Frist Treatment until 30 days after end of treatment, up to 5 months
  Rate of grade 3 or worse adverse events for anemia
Adverse events for leucopenia | Frist Treatment until 30 days after end of treatment, up to 5 months
  Rate of grade 3 or worse adverse events for leucopenia
Adverse events for thrombocytopenia | Frist Treatment until 30 days after end of treatment, up to 5 months
  Rate of grade 3 or worse adverse events for thrombocytopenia
Abnormal laboratory parameters | Frist Treatment until 30 days after end of treatment, up to 5 months
  Frequency of abnormal laboratory parameters
Progression Free Survival (PFS) | Progression free survival (PFS) is defined as the time from enrollment to the first documented evidence of disease progression or death; up to 16 months.
  Progression Free Survival (PFS) according to RECIST 1.1, Progression free survival (PFS) is defined as the time from enrollment to the first documented evidence of disease progression or death. If no information will be available for the evaluation of progression, patients will be censored at the timepoint of last tumor assessment.
Objective Response Rate (ORR) | defined as the time from enrollment up to 16 months.
  Objective response rate is defined as proportion of patients with a best overall response of complete response (CR) or partial response (PR). Tumor response will be evaluated using RECIST 1.1 criteria.
Overall survival | Overall survival (OS) is defined as the time from enrollment to the date of death from any cause.; up to 16 months.
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten O Götze, Dr., Principal Investigator — Institute of Clinical Cancer Research UCT - University Cancer Center Frankfurt
Locations (5):
- Germany (5):
  - Institute for Clinical Cancer Research Krankenhaus Nordwest, Frankfurt
  - Hamburg Hämatologisch-Onkologische Praxis Eppendorf-Facharztzentrum Eppendorf, Hamburg
  - Tagestherapiezentrum am ITM Universitätsmedizin Mannheim, Mannheim
  - Technische Universität München Klinikum Rechts der Isar, München
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goetze TO, Stein A, Lorenzen S, Habibzada T, Goekkurt E, Herhaus P, Loose M, Sookthai D, Brulin T, Ihrig K, Pauligk C, Al-Batran SE. Ramucirumab beyond progression plus TAS-102 in patients with advanced or metastatic esophagogastric adenocarcinoma, after treatment failure on a ramucirumab-based therapy. Int J Cancer. 2023 Nov 15;153(10):1726-1733. doi: 10.1002/ijc.34652. Epub 2023 Jul 16. PMID 37455496